CLINICAL TRIAL: NCT04680273
Title: A Phase I, Single Center, Open-Label, Partially Randomized, Two Part Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-GDC-9545 Following a Single Oral Dose (Part 1) and to Evaluate the Absolute Bioavailability of Oral Capsule Formulations of GDC-9545 F12 and F18 and the Relative Bioavailability of F18 Compared to F12 (Part 2) in Healthy Female Subjects of Non-Childbearing Potential
Brief Title: Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-GDC-9545 Following a Single Oral Dose (Part 1) and to Evaluate the Absolute and Relative Bioavailability of Oral Capsule Formulations of GDC-9545 (Part 2) in Healthy Female Subjects of Non-Childbearing Potential
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GP42662; 2020-004650-29 (EudraCT Number)
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — giredestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: [14C]-GDC-9545 (Experimental): Participants will be enrolled to receive a single dose of Carbon-14 labelled [14C]-GDC-9545.
  Interventions: Drug: [14C]-GDC-9545
- Part 2: GDC-9545 Treatment Sequence BCD (Experimental): Participants will be randomly allocated to one of two treatment sequences (BCD for this arm). In each treatment period, participants will receive a single dose of GDC-9545 in the fasted state in each of three treatment periods. The three treatment periods will be separated by a treatment-free washout between each study drug administration.
  Interventions: Drug: GDC-9545 Solution for Infusion; Drug: GDC-9545/F12 Capsule; Drug: GDC-9545/F18 Capsule
- Part 2: GDC-9545 Treatment Sequence BDC (Experimental): Participants will be randomly allocated to one of two treatment sequences (BDC for this arm). In each treatment period, participants will receive a single dose of GDC-9545 in the fasted state in each of three treatment periods. The three treatment periods will be separated by a treatment-free washout between each study drug administration.
  Interventions: Drug: GDC-9545 Solution for Infusion; Drug: GDC-9545/F12 Capsule; Drug: GDC-9545/F18 Capsule

INTERVENTIONS:
Drug: [14C]-GDC-9545 — Participants will receive a single oral dose of [14C]-GDC-9545 capsule, 30 milligrams (mg) (not more than [NMT] 4.6 megabecquerel [MBq]; 124 microcurie [μCi]) with approximately 240 millilitres (mL) water in the fasted state.
  Other Names: Giredestrant; RO7197597; RG6171
  Arms: Part 1: [14C]-GDC-9545
Drug: GDC-9545 Solution for Infusion — Treatment B: 30 mg GDC-9545 as a solution for infusion, 3 mg/mL administered intravenously (IV) in 10 mL as an infusion over 30 minutes.
  Other Names: Giredestrant; RO7197597; RG6171
  Arms: Part 2: GDC-9545 Treatment Sequence BCD; Part 2: GDC-9545 Treatment Sequence BDC
Drug: GDC-9545/F12 Capsule — Treatment C: GDC-9545/F12 capsule, 30 mg, administered orally with approximately 240 mL water.
  Other Names: Giredestrant; RO7197597; RG6171
  Arms: Part 2: GDC-9545 Treatment Sequence BCD; Part 2: GDC-9545 Treatment Sequence BDC
Drug: GDC-9545/F18 Capsule — Treatment D: GDC-9545/F18 capsule, 30 mg, administered orally with approximately 240 mL water.
  Other Names: Giredestrant; RO7197597; RG6171
  Arms: Part 2: GDC-9545 Treatment Sequence BCD; Part 2: GDC-9545 Treatment Sequence BDC

SUMMARY:
This is an open-label, single-center, two part study in healthy female subjects of non-childbearing potential to investigate the absorption, metabolism, and excretion of [14C]-GDC-9545 (Part 1), the absolute bioavailability of formulations F12 and F18 (i.e., GDC-9545/F12 capsule, 30 mg and GDC-9545/F18 capsule, 30 mg) and relative bioavailability of GDC-9545 oral capsule F18 to the F12 formulation (Part 2). It is planned that Part 1 will begin prior to Part 2 of the study, and that the two parts of the study will partially overlap.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non-childbearing potential that are non-pregnant, non-lactating females, who are either postmenopausal or surgically sterile, aged 30 to 65 years, inclusive, at time of signing the Informed Consent Form (ICF)
* A body mass index (BMI) between 18.5 and 32.0 kg/m^2, inclusive, at screening
* Ability to comply with the study protocol
* Must have regular bowel movements (i.e., average stool production of ≥1 and ≤3 stools per day) (Part 1 only)

Exclusion Criteria:

* Women of childbearing potential, women who are pregnant or breastfeeding
* Subjects who have received any investigational medicinal product (IMP) in a clinical research study within the 90 days prior to Day 1 (Part 1) or Day 1 of Period 1 (Part 2)
* History of serious adverse reaction or serious hypersensitivity to any drug or allergy to the study drug formulation excipients
* Subjects who are, or are immediate family members of, a study site or Sponsor employee
* Subjects who have previously been administered IMP in this study. Subjects who have taken part in Part 1 are not permitted to take part in Part 2.
* Evidence of current severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2; i.e., the virus that causes COVID-19) infection
* Positive for hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody at screening
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption >14 units per week
* A confirmed positive alcohol breath test at screening or admission
* Current smokers and those who have smoked within the last 12 months
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Confirmed positive drugs of abuse test result at screening or admission
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study (Part 1 only)
* Subjects who do not have suitable veins for multiple venipunctures/cannulation as assessed by the Investigator or delegate at screening
* Clinically significant abnormal clinical chemistry, hematology, coagulation or urinalysis as judged by the Investigator
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <70 mL/min using the Cockcroft-Gault equation
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal (GI) disease (especially peptic ulceration, GI bleeding, ulcerative colitis, Crohn's Disease or Irritable Bowel Syndrome), neurological or psychiatric disorder, as judged by the Investigator
* Presence or history of clinically significant allergy requiring treatment, as judged by the Investigator
* Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood
* Subjects who are taking, or have taken, any medication (e.g., prescription drugs, over-the-counter drugs, hormone replacement therapy [HRT], vaccines, topical medications, herbal or homeopathic remedies, nutritional supplements), other than up to 4 g of paracetamol per day, in the 14 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the Investigator.
* Subjects who are taking, or have taken, oral antibiotics within 4 weeks or IV antibiotics within 8 weeks prior to admission
* Subjects who are taking, or have taken, any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to admission
* History of GI surgery (with the exception of appendectomy unless it was performed within the previous 12 months) (Part 1 only)
* Acute diarrhea or constipation in the 7 days before the predicted Day 1. If screening occurs >7 days before the Day 1, this criterion will be determined on Day 1. Diarrhea will be defined as the passage of liquid feces and/or a stool frequency of greater than 3 times per day. Constipation will be defined as a failure to open the bowels for 3 days (Part 1 only)
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* History or presence of an abnormal ECG that is clinically significant in the Investigator's opinion, including complete left bundle branch block, second- or third-degree atrioventricular heart block, or evidence of prior myocardial infarction
* QT interval corrected through use of Fridericia's formula (QTcF) >440 msec demonstrated by at least two ECGs >30 minutes apart
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as structural heart disease (e.g., severe left ventricular systolic dysfunction, left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or long QT syndrome
* Confirmed (e.g., 2 consecutive measurements) baseline heart rate ≤50 bpm prior to enrollment
* Current treatment with medications that are well known to prolong the QT interval
* Absolute neutrophil count <1.3 x 10^9/L (1300/μL)
* Failure to satisfy the Investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: [14C]-GDC-9545: In Part 1, each participant received a single oral dose of Carbon-14 labelled [14C]-GDC-9545 capsule, 30 mg (NMT 4.6 MBq [124 μCi]). The test formulation was swallowed whole with approximately 240 mL water following an overnight fast of a minimum of 10 hours.
- Part 2: GDC-9545 Treatment Sequence BCD: In Part 2, participants were randomly allocated to one of two treatment sequences; Treatments B, C, and then D for this arm. In each of the three treatment periods, participants in the fasted state received a single 30-milligram (mg) dose of GDC-9545, administered as one of three possible formulations: Treatment B was 30-mg GDC-9545 as a solution for infusion, 3 mg/mL administered intravenously (IV) in 10 milliliters (mL) as an infusion over 30 minutes; Treatment C was a GDC-9545/F12 capsule, 30 mg, taken orally with approximately 240 mL water; and Treatment D was a GDC-9545/F18 capsule, 30 mg, taken orally with approximately 240 mL water. There was a minimum treatment-free washout period of 10 days between each study drug administration.
- Part 2: GDC-9545 Treatment Sequence BDC: In Part 2, participants were randomly allocated to one of two treatment sequences; Treatments B, D, and then C for this arm. In each of the three treatment periods, participants in the fasted state received a single 30-milligram (mg) dose of GDC-9545, administered as one of three possible formulations: Treatment B was 30-mg GDC-9545 as a solution for infusion, 3 mg/mL administered intravenously (IV) in 10 milliliters (mL) as an infusion over 30 minutes; Treatment D was a GDC-9545/F18 capsule, 30 mg, taken orally with approximately 240 mL water; and Treatment C was a GDC-9545/F12 capsule, 30 mg, taken orally with approximately 240 mL water. There was a minimum treatment-free washout period of 10 days between each study drug administration.
Period: Overall Study
Arm/Group | Part 1: [14C]-GDC-9545 | Part 2: GDC-9545 Treatment Sequence BCD | Part 2: GDC-9545 Treatment Sequence BDC
Started | 6 | 5 | 5
Part 1: Received the Planned Dose of Study Drug | 6 | 0 | 0
Part 2: Received All 3 Planned Doses of Study Drug | 0 | 5 | 5
Completed | 6 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants includes a total of 16 participants who were enrolled in either Part 1 (N = 6) or Part 2 (N = 10) of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: [14C]-GDC-9545 | Part 2: GDC-9545 Treatment Sequence BCD | Part 2: GDC-9545 Treatment Sequence BDC | Total
Number analyzed (Participants) | 6 | 5 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Baseline characteristics and results were analyzed separately for participants who were enrolled in Part 1 (N = 6) or Part 2 (N = 10) of the study.
  Years
    Part 1: number analyzed (Participants) | 6 | 0 | 0 | 6
    Part 1 | 56.2 (3.5) |  |  | 56.2 (3.5)
    Part 2: number analyzed (Participants) | 0 | 5 | 5 | 10
    Part 2 |  | 58.8 (5.6) | 57.6 (3.0) | 58.2 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics and results were analyzed separately for participants who were enrolled in Part 1 (N = 6) or Part 2 (N = 10) of the study.
  Participants
    Part 1: number analyzed (Participants) | 6 | 0 | 0 | 6
    Part 1: Female | 6 |  |  | 6
    Part 1: Male | 0 |  |  | 0
    Part 2: number analyzed (Participants) | 0 | 5 | 5 | 10
    Part 2: Female |  | 5 | 5 | 10
    Part 2: Male |  | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics and results were analyzed separately for participants who were enrolled in Part 1 (N = 6) or Part 2 (N = 10) of the study.
  Participants
    Part 1: number analyzed (Participants) | 6 | 0 | 0 | 6
    Part 1: Hispanic or Latino | 0 |  |  | 0
    Part 1: Not Hispanic or Latino | 6 |  |  | 6
    Part 1: Unknown or Not Reported | 0 |  |  | 0
    Part 2: number analyzed (Participants) | 0 | 5 | 5 | 10
    Part 2: Hispanic or Latino |  | 0 | 0 | 0
    Part 2: Not Hispanic or Latino |  | 5 | 5 | 10
    Part 2: Unknown or Not Reported |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics and results were analyzed separately for participants who were enrolled in Part 1 (N = 6) or Part 2 (N = 10) of the study.
  Participants
    Part 1: number analyzed (Participants) | 6 | 0 | 0 | 6
    Part 1: American Indian or Alaska Native | 0 |  |  | 0
    Part 1: Asian | 0 |  |  | 0
    Part 1: Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
    Part 1: Black or African American | 0 |  |  | 0
    Part 1: White | 6 |  |  | 6
    Part 1: More than one race | 0 |  |  | 0
    Part 1: Unknown or Not Reported | 0 |  |  | 0
    Part 2: number analyzed (Participants) | 0 | 5 | 5 | 10
    Part 2: American Indian or Alaska Native |  | 0 | 0 | 0
    Part 2: Asian |  | 0 | 0 | 0
    Part 2: Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0
    Part 2: Black or African American |  | 0 | 0 | 0
    Part 2: White |  | 5 | 5 | 10
    Part 2: More than one race |  | 0 | 0 | 0
    Part 2: Unknown or Not Reported |  | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Mean Cumulative Amount of Total Radioactivity (CumAe) of [14C]-GDC-9545 Excreted in Urine, Feces, and Total (Urine and Feces Combined) Over the Entire Collection Period
Description: Following a single oral dose of 30 milligrams of [14C]-GDC-9545, urine and fecal samples were collected over time from each participant. The amounts of total radioactivity excreted in the samples were determined using liquid scintillation counting. The lower limits of detection in urine and fecal samples were 0.423 and 8.36 nanogram equivalent of free drug per gram of sample, respectively. Following Day 21 (480 hours), where urine/fecal collections were no longer continuous and spot sampling days commenced, interpolation of Ae was calculated to estimate the amount excreted on non-collection days (collection intervals with interpolated values included 480-648 hours, 672-816 hours, and 840-984 hours).
Time Frame: From Day 1 to Day 42 (0-1008 hours)
Population: Mass Balance Population, Part 1: all participants who received a dose of study drug, had evaluable total radioactivity concentration (urinary and fecal) data, and had no protocol deviations that affected the mass balance analysis (e.g., spillage or missing collections, or vomiting).
Measure: Mean (Standard Deviation); unit: milligram equivalent of free drug
Groups:
- Part 1: [14C]-GDC-9545 - Urine: This analysis group represents the total radioactivity recovered from the participants' urine samples. In Part 1, each participant received a single oral dose of Carbon-14 labelled [14C]-GDC-9545 capsule, 30 mg (NMT 4.6 MBq [124 μCi]). The test formulation was swallowed whole with approximately 240 mL water following an overnight fast of a minimum of 10 hours.
- Part 1: [14C]-GDC-9545 - Feces: This analysis group represents the total radioactivity recovered from the participants' fecal samples. In Part 1, each participant received a single oral dose of Carbon-14 labelled [14C]-GDC-9545 capsule, 30 mg (NMT 4.6 MBq [124 μCi]). The test formulation was swallowed whole with approximately 240 mL water following an overnight fast of a minimum of 10 hours.
- Part 1: [14C]-GDC-9545 - Total (Urine and Feces): This analysis group represents the total radioactivity recovered from the participants' urine and feces samples combined. In Part 1, each participant received a single oral dose of Carbon-14 labelled [14C]-GDC-9545 capsule, 30 mg (NMT 4.6 MBq [124 μCi]). The test formulation was swallowed whole with approximately 240 mL water following an overnight fast of a minimum of 10 hours
Arm/Group | Part 1: [14C]-GDC-9545 - Urine | Part 1: [14C]-GDC-9545 - Feces | Part 1: [14C]-GDC-9545 - Total (Urine and Feces)
Number analyzed (Participants) | 6 | 6 | 6
milligram equivalent of free drug | 2.78 (0.503) | 20.70 (0.712) | 23.50 (0.952)

2. Primary Outcome: Part 1: Mean Cumulative Amount of Total Radioactivity Expressed as a Percentage of the Radioactive Dose Administered (CumFe) of [14C]-GDC-9545 Recovered in Urine, Feces, and Total (Urine and Feces Combined) Over the Entire Collection Period
Description: as for outcome 1
Time Frame: From Day 1 to Day 42 (0-1008 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of radioactive dose
Groups:
- Part 1: [14C]-GDC-9545 - Feces: This analysis group represents the total radioactivity recovered from the participants' feces samples. In Part 1, each participant received a single oral dose of Carbon-14 labelled [14C]-GDC-9545 capsule, 30 mg (NMT 4.6 MBq [124 μCi]). The test formulation was swallowed whole with approximately 240 mL water following an overnight fast of a minimum of 10 hours.
Arm/Group | Part 1: [14C]-GDC-9545 - Urine | Part 1: [14C]-GDC-9545 - Feces | Part 1: [14C]-GDC-9545 - Total (Urine and Feces)
Number analyzed (Participants) | 6 | 6 | 6
Percentage of radioactive dose | 9.039 (1.634) | 67.410 (2.313) | 77.012 (2.794)

3. Primary Outcome: Part 1: Mean Amount of Total Radioactivity (Ae) of [14C]-GDC-9545 Excreted in Urine, Feces, and Total (Urine and Feces Combined) by Collection Interval
Description: as for outcome 1
Time Frame: 0-12, 12-24, 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264, 264-288, 288-312, 312-336, 336-360, 360-384, 384-408, 408-432, 432-456, 456-480, 480-648, 648-672, 672-816, 816-840, 840-984, & 984-1008 hours
Population: Mass Balance Population, Part 1: all participants who received a dose of study drug, had evaluable total radioactivity concentration (urinary and fecal) data, and had no protocol deviations that affected the mass balance analysis (e.g., spillage or missing collections, or vomiting). Only urine samples were collected over 2 intervals in the first 24 hours postdose: 0-12 hours and 12-24 hours; fecal samples were collected over a single 0-24 hours interval.
Measure: Mean (Standard Deviation); unit: nanogram equivalent of free drug
Arm/Group | Part 1: [14C]-GDC-9545 - Urine | Part 1: [14C]-GDC-9545 - Feces | Part 1: [14C]-GDC-9545 - Total (Urine and Feces)
Number analyzed (Participants) | 6 | 6 | 6
nanogram equivalent of free drug
  0-12 hours: number analyzed (Participants) | 6 | 0 | 0
  0-12 hours | 668000 (78600) |  |
  12-24 hours: number analyzed (Participants) | 6 | 0 | 0
  12-24 hours | 307000 (54300) |  |
  0-24 hours: number analyzed (Participants) | 0 | 6 | 6
  0-24 hours |  | 6980 (17100) | 982000 (140000)
  24-48 hours | 410000 (56400) | 1980000 (3240000) | 2390000 (3250000)
  48-72 hours | 242000 (50600) | 3880000 (4230000) | 4120000 (4200000)
  72-96 hours | 174000 (54800) | 5730000 (4420000) | 5900000 (4380000)
  96-120 hours | 129000 (48000) | 902000 (746000) | 1030000 (761000)
  120-144 hours | 94100 (41100) | 2330000 (2590000) | 2420000 (2620000)
  144-168 hours | 56100 (22000) | 1180000 (894000) | 1240000 (905000)
  168-192 hours | 54300 (20300) | 453000 (357000) | 507000 (352000)
  192-216 hours | 49900 (21900) | 438000 (596000) | 488000 (603000)
  216-240 hours | 27700 (13600) | 732000 (1010000) | 760000 (1020000)
  240-264 hours | 35300 (13300) | 424000 (349000) | 459000 (358000)
  264-288 hours | 30000 (9410) | 470000 (633000) | 500000 (639000)
  288-312 hours | 27800 (9520) | 198000 (178000) | 226000 (187000)
  312-336 hours | 23200 (5850) | 188000 (159000) | 211000 (162000)
  336-360 hours | 25200 (4160) | 63700 (66000) | 88800 (67100)
  360-384 hours | 20300 (5510) | 159000 (68800) | 179000 (70700)
  384-408 hours | 17600 (3550) | 122000 (95300) | 139000 (96700)
  408-432 hours | 20800 (4430) | 69100 (50400) | 89900 (51200)
  432-456 hours | 17300 (2920) | 73500 (54000) | 90700 (55900)
  456-480 hours | 16300 (2940) | 82000 (45000) | 98200 (46000)
  480-648 hours | 114000 (22100) | 305000 (273000) | 401000 (161000)
  648-672 hours | 16300 (3820) | 44300 (48600) | 60600 (51700)
  672-816 hours | 93100 (19200) | 362000 (296000) | 493000 (267000)
  816-840 hours | 14700 (2830) | 88800 (70800) | 104000 (72300)
  840-984 hours | 83900 (15500) | 412000 (291000) | 496000 (300000)
  984-1008 hours | 13300 (2430) | 48500 (30200) | 61800 (32000)

4. Primary Outcome: Part 1: Mean Cumulative Amount of Total Radioactivity (CumAe) of [14C]-GDC-9545 Excreted in Urine, Feces, and Total (Urine and Feces Combined) by Cumulative Collection Interval
Description: as for outcome 1
Time Frame: 0-24, 0-48, 0-72, 0-96, 0-120, 0-144, 0-168, 0-192, 0-216, 0-240, 0-264, 0-288, 0-312, 0-336, 0-360, 0-384, 0-408, 0-432, 0-456, 0-480, 0-648, 0-672, 0-816, 0-840, 0-984, and 0-1008 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram equivalent of free drug
Arm/Group | Part 1: [14C]-GDC-9545 - Urine | Part 1: [14C]-GDC-9545 - Feces | Part 1: [14C]-GDC-9545 - Total (Urine and Feces)
Number analyzed (Participants) | 6 | 6 | 6
nanogram equivalent of free drug
  0-24 hours | 975000 (128000) | 6980 (17100) | 982000 (140000)
  0-48 hours | 1380000 (175000) | 1980000 (3230000) | 3370000 (3230000)
  0-72 hours | 1630000 (215000) | 5860000 (4840000) | 7490000 (4750000)
  0-96 hours | 1800000 (262000) | 11600000 (5790000) | 13400000 (5640000)
  0-120 hours | 1930000 (299000) | 12500000 (5520000) | 14400000 (5330000)
  0-144 hours | 2020000 (334000) | 14800000 (3120000) | 16800000 (2880000)
  0-168 hours | 2080000 (352000) | 16000000 (2740000) | 18100000 (2510000)
  0-192 hours | 2130000 (370000) | 16500000 (2840000) | 18600000 (2590000)
  0-216 hours | 2180000 (389000) | 16900000 (2650000) | 19100000 (2380000)
  0-240 hours | 2210000 (401000) | 17600000 (1820000) | 19800000 (1540000)
  0-264 hours | 2250000 (413000) | 18100000 (1620000) | 20300000 (1340000)
  0-288 hours | 2280000 (421000) | 18500000 (1280000) | 20800000 (1030000)
  0-312 hours | 2300000 (430000) | 18700000 (1160000) | 21000000 (940000)
  0-336 hours | 2330000 (436000) | 18900000 (1110000) | 21200000 (920000)
  0-360 hours | 2350000 (439000) | 19000000 (1120000) | 21300000 (932000)
  0-384 hours | 2370000 (445000) | 19100000 (1110000) | 21500000 (934000)
  0-408 hours | 2390000 (448000) | 19300000 (1060000) | 21600000 (894000)
  0-432 hours | 2410000 (451000) | 19300000 (1070000) | 21700000 (893000)
  0-456 hours | 2430000 (454000) | 19400000 (1030000) | 21800000 (854000)
  0-480 hours | 2450000 (456000) | 19500000 (1050000) | 21900000 (878000)
  0-648 hours | 2560000 (473000) | 19800000 (1010000) | 22300000 (966000)
  0-672 hours | 2580000 (475000) | 19800000 (969000) | 22400000 (922000)
  0-816 hours | 2670000 (488000) | 20200000 (742000) | 22900000 (825000)
  0-840 hours | 2680000 (490000) | 20300000 (733000) | 23000000 (847000)
  0-984 hours | 2770000 (501000) | 20700000 (719000) | 23500000 (949000)
  0-1008 hours | 2780000 (503000) | 20700000 (712000) | 23500000 (952000)

5. Primary Outcome: Part 1: Mean Amount of Total Radioactivity Expressed as a Percentage of the Radioactive Dose Administered (Fe) of [14C]-GDC-9545 Recovered in Urine, Feces, and Total (Urine and Feces Combined) by Collection Interval
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of radioactive dose
Arm/Group | Part 1: [14C]-GDC-9545 - Urine | Part 1: [14C]-GDC-9545 - Feces | Part 1: [14C]-GDC-9545 - Total (Urine and Feces)
Number analyzed (Participants) | 6 | 6 | 6
Percentage of radioactive dose
  0-12 hours: number analyzed (Participants) | 6 | 0 | 0
  0-12 hours | 2.172 (0.255) |  |
  12-24 hours: number analyzed (Participants) | 6 | 0 | 0
  12-24 hours | 0.997 (0.176) |  |
  0-24 hours: number analyzed (Participants) | 0 | 6 | 6
  0-24 hours |  | 0.023 (0.056) | 3.191 (0.454)
  24-48 hours | 1.331 (0.183) | 6.428 (10.516) | 7.759 (10.575)
  48-72 hours | 0.787 (0.164) | 12.603 (13.735) | 13.390 (13.639)
  72-96 hours | 0.566 (0.178) | 18.625 (14.351) | 19.191 (14.234)
  96-120 hours | 0.420 (0.156) | 2.932 (2.423) | 3.352 (2.472)
  120-144 hours | 0.306 (0.134) | 7.565 (8.420) | 7.871 (8.510)
  144-168 hours | 0.182 (0.072) | 3.848 (2.905) | 4.030 (2.941)
  168-192 hours | 0.176 (0.066) | 1.471 (1.159) | 1.647 (1.145)
  192-216 hours | 0.162 (0.071) | 1.424 (1.937) | 1.586 (1.961)
  216-240 hours | 0.090 (0.044) | 2.379 (3.280) | 2.469 (3.319)
  240-264 hours | 0.115 (0.043) | 1.377 (1.134) | 1.492 (1.164)
  264-288 hours | 0.098 (0.031) | 1.528 (2.056) | 1.626 (2.077)
  288-312 hours | 0.090 (0.031) | 0.644 (0.580) | 0.734 (0.608)
  312-336 hours | 0.075 (0.019) | 0.612 (0.518) | 0.687 (0.527)
  336-360 hours | 0.082 (0.014) | 0.207 (0.214) | 0.289 (0.218)
  360-384 hours | 0.066 (0.018) | 0.517 (0.224) | 0.583 (0.230)
  384-408 hours | 0.057 (0.012) | 0.396 (0.310) | 0.453 (0.314)
  408-432 hours | 0.068 (0.014) | 0.225 (0.164) | 0.292 (0.166)
  432-456 hours | 0.056 (0.009) | 0.239 (0.175) | 0.295 (0.182)
  456-480 hours | 0.053 (0.010) | 0.266 (0.146) | 0.319 (0.150)
  480-648 hours | 0.371 (0.072) | 0.993 (0.889) | 1.808 (0.518)
  648-672 hours | 0.053 (0.012) | 0.144 (0.158) | 0.197 (0.168)
  672-816 hours | 0.303 (0.062) | 1.178 (0.963) | 1.601 (0.868)
  816-840 hours | 0.048 (0.009) | 0.289 (0.230) | 0.337 (0.235)
  840-984 hours | 0.273 (0.050) | 1.339 (0.945) | 1.612 (0.974)
  984-1008 hours | 0.043 (0.008) | 0.158 (0.098) | 0.201 (0.104)

6. Primary Outcome: Part 1: Mean Cumulative Amount of Total Radioactivity Expressed as a Percentage of the Radioactive Dose Administered (CumFe) of [14C]-GDC-9545 Recovered in Urine, Feces, and Total (Urine and Feces Combined) by Cumulative Collection Interval
Description: as for outcome 1
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of radioactive dose
Arm/Group | Part 1: [14C]-GDC-9545 - Urine | Part 1: [14C]-GDC-9545 - Feces | Part 1: [14C]-GDC-9545 - Total (Urine and Feces)
Number analyzed (Participants) | 6 | 6 | 6
Percentage of radioactive dose
  0-24 hours | 3.169 (0.415) | 0.023 (0.056) | 3.191 (0.454)
  0-48 hours | 4.500 (0.570) | 6.451 (10.500) | 10.950 (10.498)
  0-72 hours | 5.286 (0.700) | 19.054 (15.718) | 24.340 (15.443)
  0-96 hours | 5.853 (0.850) | 37.679 (18.821) | 43.532 (18.320)
  0-120 hours | 6.272 (0.973) | 40.611 (17.941) | 46.884 (17.339)
  0-144 hours | 6.578 (1.086) | 48.176 (10.145) | 54.755 (9.345)
  0-168 hours | 6.761 (1.144) | 52.024 (8.919) | 58.785 (8.143)
  0-192 hours | 6.937 (1.203) | 53.495 (9.231) | 60.432 (8.410)
  0-216 hours | 7.099 (1.264) | 54.919 (8.629) | 62.018 (7.723)
  0-240 hours | 7.189 (1.303) | 57.298 (5.922) | 64.487 (4.999)
  0-264 hours | 7.304 (1.343) | 58.676 (5.269) | 65.979 (4.345)
  0-288 hours | 7.401 (1.369) | 60.204 (4.176) | 67.605 (3.358)
  0-312 hours | 7.492 (1.399) | 60.848 (3.784) | 68.339 (3.055)
  0-336 hours | 7.567 (1.416) | 61.459 (3.615) | 69.026 (2.990)
  0-360 hours | 7.649 (1.428) | 61.666 (3.645) | 69.315 (3.029)
  0-384 hours | 7.715 (1.445) | 62.183 (3.623) | 69.898 (3.035)
  0-408 hours | 7.772 (1.455) | 62.579 (3.453) | 70.351 (2.905)
  0-432 hours | 7.839 (1.467) | 62.804 (3.463) | 70.643 (2.903)
  0-456 hours | 7.895 (1.475) | 63.043 (3.346) | 70.938 (2.774)
  0-480 hours | 7.948 (1.483) | 63.309 (3.408) | 71.257 (2.853)
  0-648 hours | 8.319 (1.536) | 64.302 (3.285) | 73.065 (2.673)
  0-672 hours | 8.372 (1.543) | 64.446 (3.150) | 73.262 (2.540)
  0-816 hours | 8.675 (1.585) | 65.624 (2.412) | 74.863 (2.281)
  0-840 hours | 8.723 (1.592) | 65.913 (2.383) | 75.200 (2.365)
  0-984 hours | 8.995 (1.629) | 67.252 (2.336) | 76.812 (2.771)
  0-1008 hours | 9.039 (1.634) | 67.410 (2.313) | 77.012 (2.794)

7. Primary Outcome: Part 1: Maximum Observed Concentration (Cmax), Estimated for GDC-9545 in Plasma and for Total Radioactivity in Plasma and Whole Blood
Description: Pharmacokinetic parameters were estimated where possible and appropriate for each participant profile by non-compartmental analysis methods using Phoenix WinNonlin software. Plasma concentrations of GDC-9545 were determined using liquid chromatography with tandem mass spectrometry. Total radioactivity concentrations in plasma and whole blood were determined using liquid scintillation counting. The unit of measure for the total radioactivity concentrations is nanogram equivalent of free drug per millilitre.
Time Frame: Pre-dose and 1, 1.5, 2, 2.5, 3, 5, 6, 8, and 12 hours post-dose on Day 1, daily from Day 2 to Day 21, and Days 28, 35, and 42
Population: Pharmacokinetics (PK) Population, Part 1: all participants who received at least one dose and who satisfied the following criteria for at least one PK profile: no missing samples or invalid results at critical timepoints; no relevant protocol deviations; and, no relevant adverse events (such as vomiting).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Groups:
- Part 1: [14C]-GDC-9545 - GDC-9545 in Plasma: This analysis group represents the participants' GDC-9545 plasma samples. In Part 1, each participant received a single oral dose of Carbon-14 labelled [14C]-GDC-9545 capsule, 30 mg (NMT 4.6 MBq [124 μCi]). The test formulation was swallowed whole with approximately 240 mL water following an overnight fast of a minimum of 10 hours.
- Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma: This analysis group represents the participants' total radioactivity plasma samples. In Part 1, each participant received a single oral dose of Carbon-14 labelled [14C]-GDC-9545 capsule, 30 mg (NMT 4.6 MBq [124 μCi]). The test formulation was swallowed whole with approximately 240 mL water following an overnight fast of a minimum of 10 hours.
- Part 1: [14C]-GDC-9545 - Total Radioactivity in Whole Blood: This analysis group represents the participants' total radioactivity whole blood samples. In Part 1, each participant received a single oral dose of Carbon-14 labelled [14C]-GDC-9545 capsule, 30 mg (NMT 4.6 MBq [124 μCi]). The test formulation was swallowed whole with approximately 240 mL water following an overnight fast of a minimum of 10 hours.
Arm/Group | Part 1: [14C]-GDC-9545 - GDC-9545 in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Whole Blood
Number analyzed (Participants) | 6 | 6 | 6
nanogram per millilitre (ng/mL) | 74.3 (31.2) | 124 (21.4) | 88.0 (25.8)

8. Primary Outcome: Part 1: Time to Maximum Observed Concentration (Tmax), Estimated for GDC-9545 in Plasma and for Total Radioactivity in Plasma and Whole Blood
Description: Pharmacokinetic parameters were estimated where possible and appropriate for each participant profile by non-compartmental analysis methods using Phoenix WinNonlin software. Plasma concentrations of GDC-9545 were determined using liquid chromatography with tandem mass spectrometry. Total radioactivity concentrations in plasma and whole blood were determined using liquid scintillation counting.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: [14C]-GDC-9545 - GDC-9545 in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Whole Blood
Number analyzed (Participants) | 6 | 6 | 6
Hours | 3.50 [2.00 to 5.00] | 5.00 [2.00 to 5.00] | 5.00 [2.50 to 5.00]

9. Primary Outcome: Part 1: Area Under the Concentration-Time Curve From Time 0 to 72 Hours [AUC(0-72)], Estimated for GDC-9545 in Plasma and for Total Radioactivity in Plasma and Whole Blood
Description: as for outcome 8
Time Frame: Pre-dose and post-dose at 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, and 72 hours
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hours per milliltre (ng*h/mL)
Arm/Group | Part 1: [14C]-GDC-9545 - GDC-9545 in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Whole Blood
Number analyzed (Participants) | 6 | 6 | 6
nanogram*hours per milliltre (ng*h/mL) | 1930 (32.2) | 3370 (24.4) | 2530 (22.5)
Statistical Analysis 1: Comparison: Part 1: [14C]-GDC-9545 - GDC-9545 in Plasma vs Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma; The geometric mean ratio was calculated for the AUC(0-72) of GDC-9545 in plasma samples compared with the AUC(0-72) of total radioactivity in plasma samples; Test type: Other; Geometric mean ratio = 0.573, Standard Deviation 1.110 — The geometric coefficient of variation (%) for the AUC(0-72) geometric mean ratio was 10.4%. The standard deviation (SD) reported is a geometric SD
Statistical Analysis 2: Comparison: Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma vs Part 1: [14C]-GDC-9545 - Total Radioactivity in Whole Blood; The geometric mean ratio was calculated for the AUC(0-72) of total radioactivity (TR) in whole blood samples compared with the AUC(0-72) of TR in plasma samples; Test type: Other; Geometric mean ratio = 0.752, Standard Deviation 1.036 — The geometric coefficient of variation (%) for the AUC(0-72) geometric mean ratio was 3.5%. The standard deviation (SD) reported is a geometric SD

10. Primary Outcome: Part 1: Area Under the Concentration-Time Curve From Time 0 to the Time of Last Measurable Concentration [AUC(0-t)], Estimated for GDC-9545 in Plasma and for Total Radioactivity in Plasma and Whole Blood
Description: as for outcome 8
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hours per milliltre (ng*h/mL)
Arm/Group | Part 1: [14C]-GDC-9545 - GDC-9545 in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Whole Blood
Number analyzed (Participants) | 6 | 6 | 6
nanogram*hours per milliltre (ng*h/mL) | 2600 (43.8) | 4160 (40.3) | 3280 (40.9)
Statistical Analysis 1: Comparison: Part 1: [14C]-GDC-9545 - GDC-9545 in Plasma vs Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma; The geometric mean ratio was calculated for the AUC(0-t) of GDC-9545 in plasma samples compared with the AUC(0-t) of total radioactivity in plasma samples; Test type: Other; Geometric mean ratio = 0.625, Standard Deviation 1.134 — The geometric coefficient of variation (%) for the AUC(0-t) geometric mean ratio was 12.7%. The standard deviation (SD) reported is a geometric SD
Statistical Analysis 2: Comparison: Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma vs Part 1: [14C]-GDC-9545 - Total Radioactivity in Whole Blood; The geometric mean ratio was calculated for the AUC(0-t) of total radioactivity (TR) in whole blood samples compared with the AUC(0-t) of TR in plasma samples; Test type: Other; Geometric mean ratio = 0.790, Standard Deviation 1.171 — The geometric coefficient of variation (%) for the AUC(0-t) geometric mean ratio was 15.9%. The standard deviation (SD) reported is a geometric SD

11. Primary Outcome: Part 1: Area Under the Concentration-Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)], Estimated for GDC-9545 in Plasma and for Total Radioactivity in Plasma
Description: Pharmacokinetic parameters were estimated where possible and appropriate for each participant profile by non-compartmental analysis methods using Phoenix WinNonlin software. Plasma concentrations of GDC-9545 were determined using liquid chromatography with tandem mass spectrometry. Total radioactivity (TR) concentrations in plasma and whole blood were determined using liquid scintillation counting.
Time Frame: as for outcome 7
Population: Pharmacokinetics (PK) Population, Part 1: all participants who received at least one dose and who satisfied the following criteria for at least one PK profile: no missing samples or invalid results at critical timepoints; no relevant protocol deviations; and, no relevant adverse events (such as vomiting). 3 participants in the TR in plasma group were excluded from analysis because their parameter estimates were considered unreliable (i.e., extrapolated portion was >20% of total).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hours per milliltre (ng*h/mL)
Arm/Group | Part 1: [14C]-GDC-9545 - GDC-9545 in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma
Number analyzed (Participants) | 6 | 3
nanogram*hours per milliltre (ng*h/mL) | 2680 (43.2) | 6480 (39.2)

12. Primary Outcome: Part 1: Terminal Elimination Half-Life (t1/2), Estimated for GDC-9545 in Plasma and for Total Radioactivity in Plasma and Whole Blood
Description: as for outcome 11
Time Frame: as for outcome 7
Population: Pharmacokinetics (PK) Population, Part 1: all participants who received at least one dose and who satisfied the following criteria for at least one PK profile: no missing samples or invalid results at critical timepoints; no relevant protocol deviations; and, no relevant adverse events (such as vomiting). 3 participants in the TR in whole blood group were excluded from analysis because their parameter estimates were considered unreliable (i.e., coefficient of regression for terminal slope <0.9).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: [14C]-GDC-9545 - GDC-9545 in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Whole Blood
Number analyzed (Participants) | 6 | 6 | 3
Hours | 42.6 (24.9) | 48.4 (29.4) | 50.8 (46.4)

13. Primary Outcome: Part 1: First Order Rate Constant Associated With Terminal Portion of the Curve (λz), Estimated for GDC-9545 in Plasma and for Total Radioactivity in Plasma and Whole Blood
Description: as for outcome 8
Time Frame: as for outcome 7
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/Hours
Arm/Group | Part 1: [14C]-GDC-9545 - GDC-9545 in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Whole Blood
Number analyzed (Participants) | 6 | 6 | 3
1/Hours | 0.0163 (24.9) | 0.0143 (29.4) | 0.0136 (46.4)

14. Primary Outcome: Part 1: Total Body Clearance Calculated After a Single Extravascular Administration Where Fraction of Dose Bioavailable is Unknown (CL/F), Estimated for GDC-9545 in Plasma
Description: as for outcome 8
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres per hour (L/h)
Arm/Group | Part 1: [14C]-GDC-9545 - GDC-9545 in Plasma
Number analyzed (Participants) | 6
Litres per hour (L/h) | 11.5 (43.2)

15. Primary Outcome: Part 1: Apparent Volume of Distribution Where Fraction of Dose Bioavailable is Unknown (Vz/F), Estimated for GDC-9545 in Plasma
Description: as for outcome 8
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres per hour (L/h)
Arm/Group | Part 1: [14C]-GDC-9545 - GDC-9545 in Plasma
Number analyzed (Participants) | 6
Litres per hour (L/h) | 705 (20.6)

16. Primary Outcome: Part 1: Total Radioactivity Concentrations of [14C]-GDC-9545 in Plasma and Whole Blood at Specified Timepoints
Description: Total radioactivity concentrations in plasma and whole blood were determined using liquid scintillation counting. For calculation of the geometric mean, values reported as not detectable have been set to 0.5× the limit of detection (LOD); the LOD was 11.0 nanogram equivalent of free drug per millilitre (mL).
Time Frame: Postdose at 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalent of free drug/mL
Arm/Group | Part 1: [14C]-GDC-9545 - Total Radioactivity in Plasma | Part 1: [14C]-GDC-9545 - Total Radioactivity in Whole Blood
Number analyzed (Participants) | 6 | 6
nanogram equivalent of free drug/mL
  1 Hour | 64.7 (42.1) | 48.4 (32.9)
  1.5 Hours | 88.1 (29.2) | 66.7 (24.8)
  2 Hours | 111 (25.3) | 74.3 (26.3)
  2.5 Hours | 105 (25.1) | 76.7 (27.2)
  3 Hours | 108 (25.5) | 76.3 (24.9)
  4 Hours | 101 (22.3) | 74.4 (21.9)
  5 Hours | 123 (21.3) | 85.9 (22.3)
  6 Hours | 105 (18.9) | 70.4 (19.5)
  8 Hours | 89.1 (23.6) | 64.8 (22.2)
  12 Hours | 66.6 (22.5) | 52.3 (20.8)
  24 Hours | 45.6 (24.4) | 36.0 (26.2)
  48 Hours | 34.5 (29.5) | 24.6 (26.3)
  72 Hours | 22.7 (31.0) | 18.7 (25.0)
  96 Hours | 16.1 (64.5) | 9.97 (74.9)
  120 Hours | 9.88 (74.7) | 11.5 (64.4)
  144 Hours | 7.91 (60.3) | 7.92 (61.0)
  168 Hours | 6.64 (46.0) | 7.44 (49.2)

17. Primary Outcome: Part 1: Whole Blood to Plasma Total Radioactivity Concentration Ratios of [14C]-GDC-9545 at Specified Timepoints
Description: Total radioactivity concentrations in plasma and whole blood were determined using liquid scintillation counting. The limit of detection was 11.0 nanogram equivalent of free drug per millilitre (mL).
Time Frame: Postdose at 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours
Population: Pharmacokinetics (PK) Population, Part 1: all participants who received at least one dose and who satisfied the following criteria for at least one PK profile: no missing samples or invalid results at critical timepoints; no relevant protocol deviations; and, no relevant adverse events (such as vomiting). Participants were excluded from analysis at a given timepoint if total radioactivity was not detected in either their plasma or whole blood samples at that timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of concentrations (unitless)
Arm/Group | Part 1: [14C]-GDC-9545
Number analyzed (Participants) | 6
Ratio of concentrations (unitless)
  1 Hour | 0.747 (12.1)
  1.5 Hours | 0.758 (6.7)
  2 Hours | 0.673 (5.4)
  2.5 Hours | 0.732 (2.9)
  3 Hours | 0.704 (4.6)
  4 Hours | 0.738 (0.7)
  5 Hours | 0.700 (10.6)
  6 Hours | 0.672 (2.8)
  8 Hours | 0.728 (4.1)
  12 Hours | 0.786 (10.0)
  24 Hours | 0.789 (7.4)
  48 Hours | 0.713 (5.6)
  72 Hours | 0.825 (7.6)
  96 Hours: number analyzed (Participants) | 3
  96 Hours | 0.757 (2.0)
  120 Hours: number analyzed (Participants) | 3
  120 Hours | 1.00 (30.7)
  144 Hours: number analyzed (Participants) | 2
  144 Hours | 1.02 (27.5)
  168 Hours: number analyzed (Participants) | 1
  168 Hours | 0.843 (NA) — The geometric coefficient of variation could not be calculated with data from 1 participant.

18. Primary Outcome: Part 2: Absolute Bioavailability (F) of GDC-9545/F12 and /F18 Capsules Calculated Relative to GDC-9545 Solution for Infusion Based on the Adjusted AUC(0-∞), Estimated in Plasma Samples
Description: Absolute bioavailability of the GDC-9545/F12 and /F18 capsules were calculated relative to GDC-9545 solution for infusion based on the adjusted geometric mean AUC(0-∞) values obtained after oral and intravenous (IV) administration of GDC-9545. Log-transformed AUC(0-∞) was analyzed using mixed effects modelling techniques. The model included terms for treatment and sequence fitted as fixed effects and subject within sequence fitted as a random effect.
Time Frame: For each treatment period: Pre-dose and 0.25, 0.5, 0.58, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, and 12 hours post-dose on Day 1, and daily from Day 2 to Day 8
Population: Part 2 Pharmacokinetics (PK) Population Subset: all participants who received Treatments B and C or B and D and had reliable estimates of PK parameters for the assessment of relative bioavailability. One participant was excluded from analysis for both Treatments C and D because they did not have reliable estimates (i.e., pre-dose concentrations of GDC-9545 that were >5% of Cmax).
Measure: Geometric Mean (90% Confidence Interval); unit: Percentage
Groups:
- Part 2, PK: GDC-9545/F12 Capsule (Treatment C): This pharmacokinetics (PK) analysis set includes participants in Part 2 of the study during the treatment period in which they received a single dose of Treatment C: GDC-9545/F12 capsule, 30 mg, administered orally with approximately 240 mL water following an overnight fast of a minimum of 10 hours.
- Part 2, PK: GDC-9545/F18 Capsule (Treatment D): This pharmacokinetics (PK) analysis set includes participants in Part 2 of the study during the treatment period in which they received a single dose of Treatment D: GDC-9545/F18 capsule, 30 mg, administered orally with approximately 240 mL water following an overnight fast of a minimum of 10 hours.
Arm/Group | Part 2, PK: GDC-9545/F12 Capsule (Treatment C) | Part 2, PK: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 9 | 9
Percentage | 58.06 [53.45 to 63.07] | 58.70 [54.04 to 63.76]

19. Primary Outcome: Part 2: Relative Bioavailability Based on the Adjusted Cmax (Frel Cmax) of the GDC-9545/F18 Capsule Calculated Relative to the GDC-9545/F12 Capsule, Estimated in Plasma Samples
Description: Relative bioavailability of the GDC-9545/F18 capsule was calculated relative to the GDC-9545/F12 capsule based on the adjusted geometric mean Cmax values. Log-transformed Cmax was analyzed using mixed effects modelling techniques. The model included terms for treatment, sequence, and period fitted as fixed effects and subject nested within sequence as a random effect.
Time Frame: as for outcome 18
Population: Part 2 Pharmacokinetics (PK) Population Subset: all participants who received Treatments C and D and had reliable estimates of PK parameters for the assessment of relative bioavailability. One participant was excluded from analysis because they did not have a reliable estimate (i.e., pre-dose concentration of GDC-9545 that was >5% of Cmax).
Measure: Geometric Mean (90% Confidence Interval); unit: Percentage
Arm/Group | Part 2, PK: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 9
Percentage | 100.79 [93.87 to 108.22]

20. Primary Outcome: Part 2: Relative Bioavailability Based on the Adjusted AUC(0-∞) [Frel AUC(0-∞)] of the GDC-9545/F18 Capsule Calculated Relative to the GDC-9545/F12 Capsule, Estimated in Plasma Samples
Description: Relative bioavailability of the GDC-9545/F18 capsule was calculated relative to the GDC-9545/F12 capsule based on the adjusted geometric mean AUC(0-∞) values. Log-transformed AUC(0-∞) was analyzed using mixed effects modelling techniques. The model included terms for treatment, sequence, and period fitted as fixed effects and subject nested within sequence as a random effect.
Time Frame: as for outcome 18
Population: as for outcome 19
Measure: Geometric Mean (90% Confidence Interval); unit: Percentage
Arm/Group | Part 2, PK: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 9
Percentage | 102.04 [98.96 to 105.22]

21. Primary Outcome: Part 2: Relative Bioavailability Based on the Adjusted AUC(0-t) [Frel AUC(0-t)] of GDC-9545/F18 Capsule Calculated Relative to GDC-9545/F12 Capsule, Estimated in Plasma Samples
Description: Relative bioavailability of the GDC-9545/F18 capsule was calculated relative to the GDC-9545/F12 capsule based on the adjusted geometric mean AUC(0-t) values. Log-transformed AUC(0-t) was analyzed using mixed effects modelling techniques. The model included terms for treatment, sequence, and period fitted as fixed effects and subject nested within sequence as a random effect.
Time Frame: as for outcome 18
Population: as for outcome 19
Measure: Geometric Mean (90% Confidence Interval); unit: Percentage
Arm/Group | Part 2, PK: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 9
Percentage | 101.97 [98.44 to 105.62]

22. Secondary Outcome: Part 2: Cmax for GDC-9545 Solution for Infusion and GDC-9545/F12 and /F18 Capsules, Estimated in Plasma Samples
Description: Pharmacokinetic parameters were estimated where possible and appropriate for each participant profile by non-compartmental analysis methods using Phoenix WinNonlin software. Plasma concentrations of GDC-9545 were determined using liquid chromatography with tandem mass spectrometry.
Time Frame: as for outcome 18
Population: Pharmacokinetics (PK) Population, Part 2: all participants who received at least one dose and who satisfied the criteria for at least one PK profile. One participant was excluded from the PK analysis set for both Treatments C and D, owing to their having quantifiable pre-dose concentrations of GDC-9545 that were >5% of Cmax for both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 2, PK: GDC-9545 Solution for Infusion (Treatment B): This pharmacokinetics (PK) analysis set includes participants in Part 2 of the study who received the planned single dose of Treatment B: 30 mg GDC-9545 as a solution for infusion, 3 mg/mL administered intravenously (IV) in 10 mL as an infusion over 30 minutes following an overnight fast of a minimum of 10 hours.
Arm/Group | Part 2, PK: GDC-9545 Solution for Infusion (Treatment B) | Part 2, PK: GDC-9545/F12 Capsule (Treatment C) | Part 2, PK: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 10 | 9 | 9
ng/mL | 804 (32.3) | 94.1 (23.1) | 93.8 (31.1)

23. Secondary Outcome: Part 2: Tmax for GDC-9545 Solution for Infusion and GDC-9545/F12 and /F18 Capsules, Estimated in Plasma Samples
Description: as for outcome 22
Time Frame: as for outcome 18
Population: as for outcome 22
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2, PK: GDC-9545 Solution for Infusion (Treatment B) | Part 2, PK: GDC-9545/F12 Capsule (Treatment C) | Part 2, PK: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 10 | 9 | 9
hours | 0.50 [0.25 to 0.60] | 5.00 [2.00 to 6.00] | 4.00 [2.00 to 5.00]

24. Secondary Outcome: Part 2: AUC(0-t) for GDC-9545 Solution for Infusion and GDC-9545/F12 and /F18 Capsules, Estimated in Plasma Samples
Description: as for outcome 22
Time Frame: as for outcome 18
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part 2, PK: GDC-9545 Solution for Infusion (Treatment B) | Part 2, PK: GDC-9545/F12 Capsule (Treatment C) | Part 2, PK: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 10 | 9 | 9
ng*h/mL | 5700 (33.3) | 3120 (35.3) | 3150 (39.2)

25. Secondary Outcome: Part 2: AUC(0-∞) for GDC-9545 Solution for Infusion and GDC-9545/F12 and /F18 Capsules, Estimated in Plasma Samples
Description: as for outcome 22
Time Frame: as for outcome 18
Population: Pharmacokinetics (PK) Population, Part 2: all participants who received at least one dose and who satisfied the criteria for at least one PK profile. One participant was excluded from the PK analysis set for both Treatments C and D, owing to their having quantifiable pre-dose concentrations of GDC-9545 that were >5% of Cmax for both treatments, and 1 participant was excluded from Treatment B analysis for having an unreliable AUC(0-∞) estimate (i.e., extrapolated portion >20% of total).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part 2, PK: GDC-9545 Solution for Infusion (Treatment B) | Part 2, PK: GDC-9545/F12 Capsule (Treatment C) | Part 2, PK: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 9 | 9 | 9
ng*h/mL | 5630 (32.5) | 3270 (38.3) | 3300 (42.2)

26. Secondary Outcome: Part 2: t1/2 for GDC-9545 Solution for Infusion and GDC-9545/F12 and /F18 Capsules, Estimated in Plasma Samples
Description: as for outcome 22
Time Frame: as for outcome 18
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2, PK: GDC-9545 Solution for Infusion (Treatment B) | Part 2, PK: GDC-9545/F12 Capsule (Treatment C) | Part 2, PK: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 10 | 9 | 9
hours | 37.8 (33.9) | 35.2 (23.9) | 36.4 (21.6)

27. Secondary Outcome: Part 2: First Order Rate Constant Associated With Terminal Portion of the Curve (λz) for GDC-9545 Solution for Infusion and GDC-9545/F12 and /F18 Capsules, Estimated in Plasma Samples
Description: as for outcome 22
Time Frame: as for outcome 18
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/Hours
Arm/Group | Part 2, PK: GDC-9545 Solution for Infusion (Treatment B) | Part 2, PK: GDC-9545/F12 Capsule (Treatment C) | Part 2, PK: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 10 | 9 | 9
1/Hours | 0.0184 (33.9) | 0.0197 (23.9) | 0.0191 (21.6)

28. Secondary Outcome: Part 2: Total Body Clearance (CL) After a Single IV Administration for GDC-9545 Solution for Infusion, Estimated in Plasma Samples
Description: as for outcome 22
Time Frame: as for outcome 18
Population: Pharmacokinetics (PK) Population, Part 2: all participants who received at least one dose and who satisfied the criteria for at least one PK profile. One participant was excluded from the PK analysis set because the AUC(0-∞) estimate was considered unreliable (i.e., extrapolated portion was >20% of total).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres per hour (L/h)
Arm/Group | Part 2, PK: GDC-9545 Solution for Infusion (Treatment B)
Number analyzed (Participants) | 9
Litres per hour (L/h) | 5.31 (32.6)

29. Secondary Outcome: Part 2: Total Body Clearance Calculated After a Single Extravascular Administration Where Fraction of Dose Bioavailable is Unknown (CL/F) for GDC-9545/F12 and /F18 Capsules, Estimated in Plasma Samples
Description: as for outcome 22
Time Frame: as for outcome 18
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres per hour (L/h)
Arm/Group | Part 2, PK: GDC-9545/F12 Capsule (Treatment C) | Part 2, PK: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 9 | 9
Litres per hour (L/h) | 9.18 (38.3) | 9.08 (42.2)

30. Secondary Outcome: Part 2: Volume of Distribution Based on the Terminal Phase Calculated Using AUC(0-∞) After a Single IV Administration (Vz) for GDC-9545 Solution for Infusion, Estimated in Plasma Samples
Description: as for outcome 22
Time Frame: as for outcome 18
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres (L)
Arm/Group | Part 2, PK: GDC-9545 Solution for Infusion (Treatment B)
Number analyzed (Participants) | 9
Litres (L) | 266 (21.5)

31. Secondary Outcome: Part 2: Apparent Volume of Distribution Based on the Terminal Phase Calculated With AUC(0-∞) After a Single Extravascular Administration Where Fraction of Dose Bioavailable is Unknown (Vz/F) for GDC-9545/F12 and /F18 Capsules, Estimated in Plasma Samples
Description: as for outcome 22
Time Frame: as for outcome 18
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres (L)
Arm/Group | Part 2, PK: GDC-9545/F12 Capsule (Treatment C) | Part 2, PK: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 9 | 9
Litres (L) | 466 (20.0) | 476 (24.5)

32. Secondary Outcome: Parts 1 and 2: Number of Participants With at Least One Adverse Event, With Severity Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
Description: All adverse events (AEs) were recorded and the investigator independently assessed the seriousness and severity of each AE. AE severity was graded on a scale from 1 to 5 using the NCI-CTCAE v5.0; any events not specifically listed in the scale were defined as: Grade 1 is mild; Grade 2 is moderate; Grade 3 is severe or medically significant; Grade 4 is life-threatening; and Grade 5 is death related to an AE. AEs of special interest were: Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law; Cases of potential drug-induced kidney injury; Grade ≥3 nausea/vomiting/diarrhea; Grade ≥2 thromboembolic events; Grade ≥3 renal failure; Grade ≥3 hepatitis or elevation in ALT or AST; Grade ≥2 vaginal or uterine hemorrhage; Grade ≥2 bradycardia; Any grade of endometrial cancer; and, Suspected transmission of an infectious agent by the study drug.
Time Frame: From Baseline until end of study (up to 42 days and 35 days for Parts 1 and 2, respectively)
Population: Safety Population: all participants who received at least one dose of study drug, grouped according to the treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: GDC-9545 Solution for Infusion (Treatment B): This safety analysis set includes all participants in Part 2 of the study during the treatment period in which they received a single dose of Treatment B: 30 mg GDC-9545 as a solution for infusion, 3 mg/mL administered intravenously (IV) in 10 mL as an infusion over 30 minutes following an overnight fast of a minimum of 10 hours.
- Part 2: GDC-9545/F12 Capsule (Treatment C): This safety analysis set includes all participants in Part 2 of the study during the treatment period in which they received a single dose of Treatment C: GDC-9545/F12 capsule, 30 mg, administered orally with approximately 240 mL water following an overnight fast of a minimum of 10 hours.
- Part 2: GDC-9545/F18 Capsule (Treatment D): This safety analysis set includes all participants in Part 2 of the study during the treatment period in which they received a single dose of Treatment D: GDC-9545/F18 capsule, 30 mg, administered orally with approximately 240 mL water following an overnight fast of a minimum of 10 hours.
- Part 2: Overall: Any GDC-9545 (Treatments B, C, or D): This safety analysis set includes all participants in Part 2 who received the three planned doses of GDC-9545 (Treatments B, C, and D) and spans all three treatment periods. In Part 2 of the study, participants were randomly allocated to one of two treatment sequences: Treatments BCD or BDC. In each of the three treatment periods, participants received a single 30 mg dose of GDC-9545 in the fasted state; GDC-9545 was administered as one of three possible formulations. There was a minimum treatment-free washout period of 10 days between each study drug administration.
Arm/Group | Part 1: [14C]-GDC-9545 | Part 2: GDC-9545 Solution for Infusion (Treatment B) | Part 2: GDC-9545/F12 Capsule (Treatment C) | Part 2: GDC-9545/F18 Capsule (Treatment D) | Part 2: Overall: Any GDC-9545 (Treatments B, C, or D)
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 10
Participants
  Any Adverse Event (AE) | 3 | 5 | 3 | 4 | 9
  Serious AE | 0 | 0 | 0 | 0 | 0
  Grade 1 AE | 3 | 4 | 3 | 2 | 6
  Grade 2 AE | 0 | 1 | 0 | 2 | 3
  Grade ≥3 AE | 0 | 0 | 0 | 0 | 0
  AE Related to Study Drug | 0 | 1 | 1 | 1 | 3
  AE Leading to Withdrawal of Study Drug | 0 | 0 | 0 | 0 | 0
  AE of Special Interest | 0 | 0 | 0 | 0 | 0

33. Secondary Outcome: Parts 1 and 2: Number of Participants With at Least One Abnormality in Laboratory Safety Tests, Reported as Adverse Events
Description: Participants provided blood samples at the specified timepoints for laboratory analysis of clinical chemistry, hematology, and coagulation panels (please refer to Appendices 1 and 2 of the protocol for a complete list). Any of the laboratory test results that were outside of a parameter's normal reference range were considered abnormalities. Not every laboratory abnormality qualified as an adverse event (AE). A laboratory test result was reported as an AE if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment.
Time Frame: Part 1: Baseline and Discharge Day (up to 21 days); Part 2: Baseline, Day -1 of each of the 3 treatment periods, and Discharge Day (up to 29 days)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: [14C]-GDC-9545 | Part 2: GDC-9545 Solution for Infusion (Treatment B) | Part 2: GDC-9545/F12 Capsule (Treatment C) | Part 2: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 6 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 0

34. Secondary Outcome: Parts 1 and 2: Number of Participants With at Least One Abnormality in Vital Sign Measurements, Reported as Adverse Events
Description: Vital sign measurements included pulse rate, systolic and diastolic blood pressure while the participant was in a supine position for 5 minutes, and oral temperature. Any of the vital sign results that were outside of a parameter's normal range were considered abnormalities. Not every vital sign abnormality qualified as an adverse event (AE). A vital sign result was reported as an AE if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment.
Time Frame: Part 1: Baseline, predose and 1, 4, and 24 hours postdose, and Discharge Day (up to 21 days); Part 2: Baseline, predose and 0.5, 1, 4, and 24 hours postdose for each of the 3 treatment periods, and Discharge Day (up to 29 days)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: [14C]-GDC-9545 | Part 2: GDC-9545 Solution for Infusion (Treatment B) | Part 2: GDC-9545/F12 Capsule (Treatment C) | Part 2: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 6 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 0

35. Secondary Outcome: Parts 1 and 2: Number of Participants With at Least One Abnormality in 12-Lead Electrocardiogram Measurements, Reported as Adverse Events
Description: The 12-lead electrocardiograms (ECG) recorded measurements of heart rate, and PR, RR, QRS, uncorrected QT, and QTcF intervals. Any of the ECG parameter results that were outside of the normal range were considered abnormalities. Not every ECG abnormality qualified as an adverse event (AE). An ECG result was reported as an AE if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment.
Time Frame: Part 1: Baseline (Day 1, predose), 1, 4, and 24 hours postdose, and Discharge Day (up to 21 days); Part 2: Baseline (Day 1, predose), 0.5, 1, 4, and 24 hours postdose for each of the 3 treatment periods, and Discharge Day (up to 29 days)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: [14C]-GDC-9545 | Part 2: GDC-9545 Solution for Infusion (Treatment B) | Part 2: GDC-9545/F12 Capsule (Treatment C) | Part 2: GDC-9545/F18 Capsule (Treatment D)
Number analyzed (Participants) | 6 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline until end of study (up to 42 days and 35 days for Parts 1 and 2, respectively)
Arm/Group | Part 1: [14C]-GDC-9545 | Part 2: GDC-9545 Solution for Infusion (Treatment B) | Part 2: GDC-9545/F12 Capsule (Treatment C) | Part 2: GDC-9545/F18 Capsule (Treatment D) | Part 2: Overall: Any GDC-9545 (Treatments B, C, or D)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/6 | 5/10 | 3/10 | 4/10 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: [14C]-GDC-9545 (N=6) | Part 2: GDC-9545 Solution for Infusion (Treatment B) (N=10) | Part 2: GDC-9545/F12 Capsule (Treatment C) (N=10) | Part 2: GDC-9545/F18 Capsule (Treatment D) (N=10) | Part 2: Overall: Any GDC-9545 (Treatments B, C, or D) (N=10)
External ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT04680273/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT04680273/SAP_001.pdf